CLINICAL TRIAL: NCT03027102
Title: Phase I Study of Allogeneic Double Negative T Cells (DNT-UHN-1) in Patients With High Risk Acute Myeloid Leukemia
Brief Title: Study of Allogeneic Double Negative T Cells (DNT-UHN-1) in Patients With High Risk Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OZM-079
Record Dates: First submitted 2017-01-04; First posted 2017-01-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: allogenic double negative T cells; DNT cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Arm (Experimental): Patients will receive DNT cells from healthy donors.
  Interventions: Biological: DNT cells
- Donor Arm (No Intervention): Healthy volunteer donors will donate blood.

INTERVENTIONS:
Biological: DNT cells — DNT cells will be expanded (increased in numbers) in the laboratory, in order to enhance their tumour destroying potential before infusion into AML patients.
  Arms: Patient Arm

SUMMARY:
This study aims to determine the safety and toxicity of incremental doses of Double Negative T (DNT) cells in human subjects with high risk acute myeloid leukemia (AML). DNT cells are mature T lymphocytes that comprise ~1% of white blood cells in humans. Injection of DNTs from healthy donors has been demonstrated to be effective against AML cells. DNT cells will be collected from healthy volunteers and injected into patients.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patients with AML who are 18 years of age or older.
2. Viably frozen cells from the time of diagnosis or relapse are available for sensitivity testing to DNT cells.
3. Patients have given informed consent.
4. Patients in remission following FLAG-Ida induction therapy who are receiving consolidation treatment.
5. Creatinine < 1.5 x ULN within 7 days prior to day 1 of study treatment.
6. AST, ALP, bilirubin < 1.5x ULN within 7 days prior to day 1 of study treatment.
7. Female patients of childbearing potential should be willing to use 2 methods of birth control (Refer to section 9.2.15 or be surgically sterile, or abstain from heterosexual activity for the course of the study from day 1 until 1 months following chemotherapy. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 years.

   Male patients should use condoms or abstain from sex from the time of beginning chemotherapy to 1 month after the chemotherapy.
8. Patients must be able to comply with study procedures, at the minimum, until all DNT-UHN-1 cells are out of their system.

Patient Exclusion Criteria:

1. ECOG performance status <2.
2. Patients with a known persistent infection.
3. Patients with known active CNS disease.
4. Life expectancy < 3 months.
5. Patients should be off Cox2 inhibitors and corticosteroids for at least 3 days prior to and 7 days after infusion of DNT cells.
6. Patients who are HIV positive.
7. Patients for whom healthy donor DNT kill <10% of patient's blast cells.

Donor Inclusion Criteria:

1. Has given written informed consent.
2. Is 18 years of age or older.
3. No known prior blood product transfusion or surgery.
4. Blood electrolytes (Sodium, Potassium, Chloride, Bicarbonate, Magnesium, Phosphate, Calcium) within normal ranges.
5. Normal complete blood counts.
6. Normal liver and kidney function (Bilirubin, AST, ALT, ALP, LDH, plasma albumin, creatinine).
7. Negative for transfusion transmissible illnesses (CMV, HIV I/II, HTLV I/II, Hepatitis B Surface Antigen, Hepatitis B Surface Antibody, Hepatitis B Core Antibody, Hepatitis C Antibody) within 30 days of blood collection for DNT cell expansion for patient infusion.
8. Negative for evidence of exposure to West Nile Virus, Syphilis within 30 days of blood collection for DNT cell expansion for patient infusion.
9. DNT cell expansion yield is >108 per mL blood using the standard protocol. Expanded DNT cells show ≥20% cytotoxicity to at least 3 AML cell lines (MV4-11 AML3, and U937).
10. The donor who meet all donor inclusion/exclusion criteria, whose DNT cells show the most potent killing (minimum >10% killing) of AML patient's blast cells (blast cells frozen at time of diagnosis or relapse) will be approached for participation in this study.

Donor Exclusion Criteria:

1. With a history of high risk behavior including, but not limited to, a history of piercing (except ear lobes), tattoos or other body modification.
2. Has serious illnesses such as cardiovascular disease & cancer.
3. Has sexually transmissible disease.
4. Has history of intravenous drug use.
5. Persons who received any vaccinations in past 3 months prior to enrolment into this study.
6. Persons who travel outside the U.S. and Canada in the past 3 years prior to enrolment into this study, to areas that are considered endemic for malaria.
7. Persons who have received blood components or other human tissues in the past 12 months prior to enrolment into this study (however this may be reduced to 6 months if nucleic acid testing (NAT) is used for the tests).
8. Pregnant or lactating.
9. Persons at risk of transmitting a hematological or immunological disease.
10. Persons with transmissible genetic diseases in the family.
11. On prescription medication.
12. Persons with prion-related disease.
13. Persons with a neurological disease of an unestablished etiology.
14. Persons with active encephalitis or meningitis of infectious or unknown etiology.
15. Persons with rabies or persons who, within the past 6 months, were bitten by an animal and treated as if the animal was rabid.
16. Persons with a family history of Creutzfeldt-Jakob disease.
17. Persons who have received human-derived pituitary growth hormone or dura mata.
18. Persons who have known or suspected sepsis at the time of donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events and abnormal laboratory studies. | 2 years
  Patients will be assessed for adverse events based upon, but not limited to, monitoring of vital signs and prescribed laboratory studies. Adverse events (AE) will use the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE). This study will utilize the CTCAE Version 4.03 for adverse event reporting.

SECONDARY OUTCOMES:
Number of cells with disease specific mutations per patient | 2 years
  Quantitive real time polymerase chain reaction (PCR) analysis for disease specific mutations will be performed on the bone marrow aspirate.
Leukemia load | 2 years
  Peripheral blood will be obtained after DNT cell infusion to monitor leukemia load and residual disease by determining the frequency of leukemic cell markers on cells using flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada